CLINICAL TRIAL: NCT03327480
Title: The Effects of Hand Orthosis in Thumb Osteoarthritis
Brief Title: The Effects of Two Different Orthosis on Pain, Hand Strength and Function in Patients With Thumb Carpometacarpal Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Aslı Can, medical doctor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aslı Can
Record Dates: First submitted 2017-10-14; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis Thumb
Keywords: osteoarthritis thumb; orthosis; functioning
MeSH Terms: interventions — Orthotic Devices

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoprene CMC orthosis (Experimental): We will prescribe a neopren CMC orthosis for patients in Group 1 and a thermoplastic CMC orthosis for patients in Group 2
  Interventions: Other: orthosis
- thermoplastic CMC orthosis (Experimental): We will prescribe a neoprene CMC orthosis for patients in Group 1 and a thermoplastic CMC orthosis for patients in Group 2
  Interventions: Other: orthosis

INTERVENTIONS:
Other: orthosis — Group 1: neoprebe CMC orthosis Group2: thermoplastic CMC orthosis

SUMMARY:
The investigators aimed to assess the effects of two different hand orthosis on hand functioning, pain, disability and quality of life in patients with thumb osteoarthritis

DETAILED DESCRIPTION:
The investigators will randomized 60 patients with stage 1 or 2 thumb osteoarthritis in two groups. The investigators will prescribe a neoprene CMC orthosis for patients in Group 1 and a thermoplastic CMC orthosis for patients in Group 2. The investigators will recommend these orthosis for six weeks. They will assess pain and disability before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 18 and 70
* Grade 1 or 2 thumb osteoarthritis

Exclusion Criteria:

* The other hand disorders such as fracture and carpal tunnel syndrome
* Previous hand surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
AUSCAN (Australian Canadian Oateoarthritis Hand Index) | before the treatment, end of the sixth week
  This scale is used to assess of pain, disability and stiffness. Change is being assesed. Total score is ranged between 0-90.